CLINICAL TRIAL: NCT03277118
Title: Quantifying Activity After Cardiac Surgery Using Wireless Wearable Technology
Brief Title: Quantifying Activity Using Wireless Wearable Technology
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sreekanth Cheruku, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 032017-102
Record Dates: First submitted 2017-05-17; First posted 2017-09-08 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Activity, Motor; Sleep; Delirium
MeSH Terms: conditions — Motor Activity; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Cohort: Patients aged 18 years or older who are scheduled to undergo elective cardiac surgery with cardiopulmonary bypass.
  Interventions: Device: Wireless Wearable Device

INTERVENTIONS:
Device: Wireless Wearable Device — Wireless Wearable Device will be placed on the wrist of the patient prior to extubation in the ICU to record patient activity in terms of steps and sleep quality.

SUMMARY:
Wireless wearable devices (WWD) have been shown to be an effective means to measure patient activity and sleep-wake cycles in the ICU. However, no current studies involving WWD have demonstrated the ability of these devices to measure adverse outcomes, including delirium in critically ill patients. This study is unique because the investigators will implement monitoring with the WWD prior to extubation in the ICU to correctly measure first mobilization, as well as capture quality of sleep and episodes of delirium for the first five postoperative days.

DETAILED DESCRIPTION:
In this single-center non-randomized prospective cohort study, cardiac surgical patients undergoing cardiac surgery with cardiopulmonary bypass will be enrolled consecutively with written informed consent from the time this protocol is approved by the IRB until 100 subjects are enrolled (expected duration of subject enrollment is 12 months). Upon arrival into the ICU, cardiac surgery subjects will have a Fitbit Charge 2 device placed on their wrist and will wear the device until the fifth post-operative day. This device will wirelessly transmit data regarding activity and sleep quality to a smartphone application for the duration of wear. No identifiable patient information will be entered into the smartphone application or transmitted to any external entity.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Adult (Age > 18) patients undergoing scheduled, elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Those who do not meet the inclusion criteria, pregnant women, prisoners, those with skin or systemic infections, those who are paraplegic or quadriplegic and those with allergies to the polyurethane material comprising the FitBit strap.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who are scheduled to undergo elective cardiac surgery at UT Southwestern Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Number of steps walked | Postoperative day 2 to Postoperative day 5
  Number of steps walked as measured by the Wireless Wearable Device

SECONDARY OUTCOMES:
Length of sleep | Postoperative Day 1
  Number of hours slept with little activity as measured by the Wireless Wearable Device
Delirium | Postoperative Day 2 (after extubation)
  Occurrence of delirium with few hours slept as measured by the Wireless Wearable Device

CONTACTS AND LOCATIONS:
Overall Officials: Sreekanth Cheruku, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No